CLINICAL TRIAL: NCT05313698
Title: Validity and Reliability of The Turkish Version of The Kidscreen-27 Questionnaires in Individuals With Cerebral Palsy
Brief Title: Validity and Reliability of The Turkish Version of The Kidscreen-27
Status: Completed | Type: Observational
Sponsor: Muş Alparslan University (Other)
Responsible Party: Principal Investigator, Hasan Bingöl, Dr, Muş Alparslan University
Other Study IDs: 16969557-2167
Record Dates: First submitted 2022-03-22; First posted 2022-04-06 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2022-05

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: No intervention — cross-sectional study/psychometric study

SUMMARY:
Functional impairment of the upper extremities can impair the health-related quality of life (HRQOL) of persons with Cerebral Palsy CP. Health-related quality of life (HRQOL) measures several subjective dimensions dealing with the impact of health or illness on physical and psychosocial functioning. Quality of life (QOL) measures for children and adolescents have been developed in recent years, initially for children with specific chronic conditions, but more recently generic and health-related QOL (HRQOL) measures have been developed . The early assessments of children's quality of life were mostly disease-specific, and this trend has continued. Generic HRQOL measurements for children and adolescents can help identify subgroups of children and adolescents who are at risk of developing health problems. KIDSCREEN-27 is a generic HRQOL measure derived from KIDSCREEN-52. The KIDSCREEN-27 is a subset of the KIDSCREEN-52 that includes 27 items for assessing HRQOL across five dimensions: Physical Well-Being (5 items) examines a child's or adolescent's level of physical activity, energy, and fitness. Although the psychometric properties of the Turkish version of the KIDSCREEN forms have been studied previously; however, its psychometric characteristics in children with CP have yet to be determined. Accordingly, the aim of this study is to provide an overview of the psychometric results of the KIDSCREEN-27 HRQOL questionnaire

DETAILED DESCRIPTION:
Children with CP generally report a lower QOL than their normally developing peers. Quality of life (QOL) is now recognized as an important outcome of interventions because it relates to a person's individual cognition or well-being in a range of domains (e.g., physical, social, emotional, spiritual). Health-related quality of life (HRQOL) is a subdomain of the more global construct of QOL, including domains such as physical, mental, and social well-being Recently, there has been a surge in interest in assessing the quality of life (QOL) of children with cerebral palsy (CP). QOL instruments are increasingly used to assess the effectiveness of interventions for children with CP. To assess QOL, there are both generic and condition-specific scales available. The Cerebral Palsy Quality of Life Questionnaire for Children (CP QOL-Child), the Child Health Questionnaire (CHQ), European generic health related quality of life questionnaire (KIDSCREEN), and the Pediatric Quality of Life Inventory are some of the most used instruments. Out of these QOL instruments, European generic health related quality of life questionnaire (KIDSCREEN) is a generic QOL questionnaire and KIDSCREEN-27 is a shorter version of the KIDSCREEN-52 questionnaire to evaluate HRQOL outcomes of children and adolescents between the ages of 8-18 years. . Generic scales are useful for comparing groups since they are designed to be relevant to all subgroups of the population. Because they do not include domains that are relevant to the sickness or disability, they are less useful for evaluating the effectiveness of an intervention for children with that illness or disability. Condition-specific scales are useful for detecting changes in QOL for a given condition and are designed to be applicable to a group. Instruments that are condition-specific can capture the domains of QOL that are significant to children and adolescents with CP. Although the psychometric properties of KIDSCREEN-27 tests have been extensively studied in healthy children and adolescents, there has been no research to date on the psychometric features of KIDSCREEN-27 instruments in cerebral palsy children and adolescents. Thus, the aims of this study were to examine and determine the construct-concurrent validity and reliability of the Turkish version of the self and proxy versions of KIDSCREEN-27 questionnaire in individuals with cerebral palsy

ELIGIBILITY:
Inclusion Criteria:

Children with cerebral palsy who have sufficient intellectual level to answer KIDSCREEN-27' items

Exclusion Criteria:

children with severe intellectual disability

Ages: 8 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Children with all typologies of cerebral palsy and their parents/caregivers
Sampling Method: Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Consistency from baseline in mean scores of KIDSCREEN-27 at week 2 | Change from Baseline KIDCREEN-27 mean scores at 2 weeks
  The KIDSCREEN-27 is a 27-item variation of the KIDSCREEN-52 questionnaire that includes five dimensions of health-related quality of life (HRQOL). It is a valid and reliable tool for assessing children's and adolescents' HRQOL outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Mintaze KEREM GUNLE, Study Chair — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)